CLINICAL TRIAL: NCT03914170
Title: A Retrospective Study Assessing the Efficacy and Safety of Triplet Chemotherapy (FOLFIRINOX) Fluorouracil + Oxaliplatin + Irinotecan Plus Cetuximab (ERBITUX®) as First Line Treatment in a RAS (Ras Sarcoma Viral Oncogene Homolog) (KRAS, NRAS) Wild-type Metastatic Colorectal Cancer Population According to BRAF (Murine Sarcoma Viral Oncogene Homolog B) Status and Primary Tumor Location
Brief Title: Folfirinox + Cetuximab Chemotherapy, in First Line, With Wild RAS and According to BRAF Status in Metastatic Colorectal Cancer
Acronym: ESTER
Status: Completed | Type: Observational
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Collaborators: Merck Serono International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: ICM-URC2016/31
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; first line; folfirinox + cetuximab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — folfirinox; Cetuximab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Folfirinox + cetuximab — Cetuximab 250 mg/m² iv infusion for 2h, Oxaliplatin 85 mg/m² administered as an iv infusion for 2h Elvorine 200 mg/m² administered as an iv infusion for 2h, Irinotecan 180 mg/m² iv infusion, 5FU 400 mg/m2 bolus then 5FU 2,400 mg/m² iv infusion for 46h D1=D15 (12 cycles max)

SUMMARY:
This retrospective study, will evaluate patient outcomes after triplet chemotherapy (FOLFIRINOX) (5 Fluorouracil + oxaliplatin + irinotecan) plus cetuximab 1st line treatment focusing on efficacy and safety in a RAS (KRAS, NRAS (neuroblastoma rat sarcoma viral oncogene homolog) wild-type metastatic colorectal cancer population, and according to BRAF (murine sarcoma viral oncogene homolog B) status and primary tumor location.

DETAILED DESCRIPTION:
In Europe, there are 447,000 new cases of colorectal cancer each year. Approximately 25% of patients present with metastases at initial diagnosis and almost 50% of patients with mCRC (metastatic colorectal cancer) will develop metastases

. Chemotherapy represents the backbone of treatment, and survival is linked with the administration of all three active cytotoxic agents (5-fluorouracil/folinate, oxaliplatin, and irinotecan) in the first line treatment of metastatic colorectal disease.

Monoclonal antibodies such as cetuximab in combination with chemotherapy are a first line treatment option in metastatic RAS (rat sarcoma viral oncogene homolog) wild type metastatic colorectal cancer (mCRC).

Phase II trials evaluating triplet chemotherapy plus cetuximab reported interesting results in terms of efficacy (response rate, resectability...), but at the price of an increased rate of toxic effects.

This retrospective study, will evaluate patient outcomes after triplet chemotherapy (FOLFIRINOX) (5 Fluorouracil + oxaliplatin + irinotecan) plus cetuximab 1st line treatment focusing on efficacy and safety in a RAS (KRAS, NRAS (neuroblastoma rat sarcoma viral oncogene homolog) wild-type mCRC (metastatic colorectal cancer) population, and according to BRAF (murine sarcoma viral oncogene homolog B) status and primary tumor location.

ELIGIBILITY:
Inclusion Criteria:

1. Colorectal cancer confirmed as RAS wild by tumor tissue analysis
2. Non resectable and measurable metastatic disease
3. Patients treated with FOLFIRINOX + cetuximab in first line metastatic disease
4. Males or females aged over 18 years.

Exclusion Criteria:

1. Known brain metastases
2. RAS not assessable (e.g., material not available or insufficient)
3. The first administration of cetuximab was more than 30 days after the first administration of FOLFIRINOX
4. History of other malignancy in the last 5 years. Patients with prior history of in situ cancer or basal or squamous cell skin cancer are eligible. Patients with other malignancies are eligible if they were cured by surgery alone or surgery plus radiotherapy and have been continuously disease-free for at least 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received FOLFIRINOX plus cetuximab (Erbitux®) in first line metastatic colorectal cancer, identified in 3 studies and Medical files from ICM in France:
  * Medical files from ICM (Montpellier)
  * UNICANCER- PRODIGE 14 study
  * ERBIRINOX study
  * EREBUS study
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Median Progression free survival (PFS) | Approximately 36 months
  In RAS wt population

SECONDARY OUTCOMES:
Progression free survival (PFS) | 9 months
  Rates in RAS wt population
Overall Response Rate | Maximal 6 months
  at the end of 1st line treatment evaluated according RECIST ( Response Evaluation Criteria in Solid Tumours)
Overall Survival | Approximately 36 months
  Defined as the time from the date of initial first line treatment initiation to the date of documented death from any cause
Duration of response | Approximately 36 months
Assessment of adverse events by using the NCI-CTCAE version 4.0 scale | Maximal 6 months
  Maximum grade observed throughout the treatment
Liver metastases resection rate | Maximal 6 months
  Resection (R0 / R1 / R2)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle SAMALIN, MD, Principal Investigator — Institut régional du cancer de Montpellier
Locations (1):
- Institut régional du cancer de Montpellier, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: No